CLINICAL TRIAL: NCT05913934
Title: Control Gait Analysis in Clubfoot Children and Comparison With Their Healthy Twins
Brief Title: Clubfeet and Twins and Gait Analysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr.Joller BioMedical Consulting (Other)
Responsible Party: Sponsor
Other Study IDs: ID 2023-00290
Record Dates: First submitted 2023-05-19; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Clubfoot
Keywords: Clubfoot; gait analysis; twin comparison; inertial sensor; footscan; manual-dynamic physiotherapy; derotation
MeSH Terms: conditions — Clubfoot | interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gait analysis parameters: Twins: Gait analysis
  Interventions: Behavioral: Gait analysis

INTERVENTIONS:
Behavioral: Gait analysis — Walk over 25 meters in a gym (GaitUp) Walk over 6 meters with footscan v9 in the office

SUMMARY:
Children with clubfeet who were exclusively treated by Ursula Issler-Wüthrich for 3 to 14 years with manual-dynamic physiotherapy and their healthy twin siblings are compared using gait analysis.

GaitUp sensors (kinematic) and footscan V9 (kinetic) are the systems used for this comparison.

Nonparametric statistics are applied to verify aberrations.

DETAILED DESCRIPTION:
Control gait analysis in clubfoot children and comparison with their healthy twins

Clubfeet are the most common birth defect with about 80 cases in Switzerland per year. There are two important therapies: Ponseti and manual-dynamic physiotherapy.

Ursula Issler-Wüthrich, physiotherapist, since twenty years treats exclusively clubfeet and comorbidities with clubfeet like arthrogryposis and myelomeningocele. Until today she corrected more than 400 feet with manual-dynamic physiotherapy.

Among her patients there are 11 twin pairs. In the scientific literature it is stated that in unilateral clubfoot, the other foot cannot be considered normal.With the two gait analysis systems meant for controlling the therapy results, the walking pattern of the healthy twin was compared with the pattern of the affected twin sibling.

The basis of the study is a walk over 25 meters with the GaitUp sensors (11 g) resulting in 22 quantitative digital parameters and tests on the pedobarographic plate footscan V9 leading to 10 parameters.

Statistically it will be analyzed whether there is a discrepancy between the clubfeet children and their healthy twins.

The parents in writing and the children orally gladly approved the task.

ELIGIBILITY:
Inclusion Criteria:

* Twins with clubfeet

Exclusion Criteria:

* All other clubfeet

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children from 3 to 14 years old, beeing treated for clubfeet and their healthy twins.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-04-29 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Differences in gait analyses of treated clubfeet and their healthy twin siblings: p-value | 2 years
  The gait analyses parameters are statistically compared between the healhy siblings and the clubfoot twins. The p-values descibe the disparity among the groups. p-values below 0.05 point to a statistical difference and are a clue to insufficient therapy.
Differences in gait analyses of treated clubfeet and their healthy twin siblings:Effect size | 2 years
  The effect size is a measure for the interpretation of differences. It represents the shift between the standard curves of the two populations. Effect sizes of more than ±0.5 suggests a serious discrepancy.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Joller, PhD, Study Director — Dr.Joller BioMedical Consulting
Locations (1):
- Dr.Joller BioMedical Consulting, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes